CLINICAL TRIAL: NCT06788353
Title: Prospective Collection of Therapeutic Efficacy and Safety Data in Patients with Unresectable Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Wei Peng, Professor, Sun Yat-sen University
Other Study IDs: [2023]546
Record Dates: First submitted 2025-01-19; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Transarterial Chemoembolization; Systemic Therapy; Unresectable Hepatocellular Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TACE alone: TACE with either cTACE or DEB-TACE can be used, depending on the selection of the patient and the physician.
- TACE plus systemic therapy: TACE with either cTACE or DEB-TACE can be used, depending on the selection of the patient and the physician.
  Systemic therapy includes target therapies and immunotherapies. Monotherapy and the combined therapy can be used, depending on the selection of the patient and the physician.

SUMMARY:
The malignant degree of middle and advanced liver cancer is very high, and the survival prognosis of patients is very poor. TACE is currently the standard treatment for unresectable liver cancer recommended by several international authoritative guidelines. However, TACE can only extend survival from 8 months to 13 months, and the prognosis for patients with unresectable liver cancer is still not optimistic. In recent years, some studies have suggested that the combination of TACE and systemic therapy can prolong OS and PFS, but a number of prospective studies have found that the combination of TACE and targeted therapy can not improve the prognosis of unresectable liver cancer. However, TACE as a non-radical treatment is difficult to achieve complete tumor necrosis, so it is still unknown which treatment combination can best improve the prognosis. This trial is an observational clinical trial to explore the efficacy and safety of TACE combined targeting/immunotherapy for unresectable hepatocellular carcinoma. Clinical data of patients with unresectable liver cancer treated in our hospital from March 2023 to March 2025 are intended to be collected to evaluate the efficacy and safety of TACE combined with different systems for unresectable liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1, age 18-75 years old; 2. Patients with primary unresectable liver cancer who have not received any previous treatment (in accordance with the AASLD 2018/EASL 2018 Liver Cancer Diagnostic guidelines); Or patients with unresectable liver cancer who recurred for the first time after radical therapy and did not receive any postoperative adjuvant therapy; 3. There is at least one lesion in the liver that can be measured according to mRECIST criteria, and the intrahepatic lesion is a single tumor ≤10.0cm or multiple tumors (the number of tumors ≤10) and the tumor load is less than 50% (three-dimensional reconstruction of CT scan using Vitelacore software [version: 6.9.87.1, Canon], calculated as proportion of tumor volume to total liver volume) 4. Normal liver tissue volume exceeds 700ml 5, ECOG score 0-1, good general condition 6, liver function Child-Pugh grade A 7. Expected survival time ≥3 months 8. Blood, liver and kidney function meet the following conditions: a) Neutrophil count ≥1.5×109/L b) Platelet count ≥60×109/L c) Hemoglobin concentration ≥90g/L d) Serum albumin concentration ≥30g/L e) bilirubin ≤50umol/L f) AST and ALT were 5 times lower than the upper limit of normal, ALP less than 4 times the upper limit of normal g) prothrombin time less than 6 seconds above the upper limit of normal h) creatinine less than 1.5 times the upper limit of normal

Exclusion Criteria:

1. Preoperative imaging examination assessed tumor load >50%;
2. Previous history of hepatic encephalopathy, refractory ascites, or esophageal and gastric varices rupture bleeding;
3. There are contraindications for TACE treatment, such as portal shunt, isolated hepatic blood flow, and obvious atherosclerosis;
4. Patients with extrahepatic metastasis;
5. Allergic to intravenous contrast agents;
6. Pregnant or lactating women or subjects who plan to have a family within two years; 7, accompanied by HIV, syphilis infection;

8. Accompanied by other malignant tumors or had other malignant tumors within 5 years prior to enrollment; 9. Allogeneic organ transplants; 10, serious heart, kidney and other organ dysfunction; 11. Active clinical severe infection > Grade 2; 12. Suffering from mental illness may affect informed consent; 13, can not take oral medicine; 14. Participated in other drug clinical trials within 12 months before enrollment; 15. Active gastric or duodenal ulcer occurred 3 months before enrollment; 16. Previous history of liver or adjacent tissue radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study populations in this study are patients with primary unresectable liver cancer who have not received any previous treatment or patients with unresectable liver cancer who recurred for the first time after radical therapy and did not receive any postoperative adjuvant therapy;
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 24 months
  Defined as the time from commencement of enrollment to progression of disease or death throughout the trial. Patients who withdraw or are lost to follow-ups will be treated as censored data, and the last date of known living without progression will be used as the last survival time. Patients whose diseases have not progressed at ending of this study will be treated as censored data, and the last date of known living without progression will be used as the last survival time.

SECONDARY OUTCOMES:
Overall survival | 24 months
  Defined as the time from the commencement of enrollment to all-cause death throughout the trial. Patients who withdraw or are lost to follow-ups will be treated as censored data, and the last date of known living will be used as the last survival time. Patients who still survive at ending of this study will also be treated as censored data, and the last date of known living is used as the last survival time.
tumor response | 24 months
  tumor response is evaluated based on mRECIST and RECIST v1.1 criteria, including complete response, partial response, stable disease, and progression disease.
Safety | 24 months
  Defined as one of ≥ grade 3 hematologic or non-hematologic toxicity events. The severity of adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE v5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiiated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No